CLINICAL TRIAL: NCT00718380
Title: An Open Label, Phase I Study Evaluating Pharmacokinetics, Safety, and Tolerability of ABT-869 in Subjects With Solid Tumors
Brief Title: A Phase 1 Study of ABT-869 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-227
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2012-07

CONDITIONS: Solid Tumor
MeSH Terms: interventions — linifanib

ARMS (4):
- Group 1 (Experimental): Dose escalation from Open label 0.05 to 0.25 mg/kg once a day dosing for 21 days
  Interventions: Drug: ABT-869
- Group 2 (Experimental): Open label 0.10 mg/kg once a day dosing after safety evolution of Group 1
  Interventions: Drug: ABT-869
- Group 3 (Experimental): Open label 0.20 mg/kg once a day dosing after safety evolution of Group 2
  Interventions: Drug: ABT-869
- Group 4 (Experimental): Open label 0.25 mg/kg once a day dosing after safety evolution of Group 3
  Interventions: Drug: ABT-869

INTERVENTIONS:
Drug: ABT-869 — 2.5 mg or 10 mg tablet, Once a day, oral dose, dose per body weight (dose determined by group; 2.5mg or 10mg tablet) until evidence of uncontrolled unacceptable toxicity or disease progression. For more information, please see Arm Description.

SUMMARY:
The objective of this study is to evaluate the pharmacokinetics, safety and tolerability of ABT-869 in Japanese patients with solid tumors up to the Recommended Phase Two Dose that was determined in a previous the M04-710 study.

ELIGIBILITY:
Inclusion Criteria

* Subjects aged from 20 to 75 years and ECOG PS of 0-2 at screening.
* Subject must have a solid tumor that is refractory to standard therapies or for which a standard effective therapy does not exist.
* The subject must have adequate bone marrow, renal and hepatic function.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation and up to six months following completion of therapy.
* The subject must voluntarily sign and date an informed consent.

Exclusion Criteria

* The subject currently exhibits symptomatic or intervention indicated CNS metastasis.
* The subject has received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic or any investigational therapy within 4 weeks of enrollment or has not fully recovered from toxicity resulting from past treatment(s) that affects the assessments in this study at the enrollment.
* The subject with the following conditions during screening assessment.

  1. proteinuria CTC grade > 1 as measured by urinalysis and 24 hour urine collection
  2. diastolic blood pressure (BP) > 95 mmHg; or systolic blood pressure (BP) > 150 mmHg
  3. a history of or currently exhibits clinically significant cancer related events of bleeding
  4. LV Ejection Fraction < 50%
  5. received a cumulative dose of Anthracycline > 360 mg/m2 for treatment of cancer
  6. receiving therapeutic anticoagulation therapy
  7. having fractures except for chronic bone lesion due to bone metastases
* The subject exhibits evidence of other clinically significant uncontrolled condition(s).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety tolerability assessment | Weekly assessment for 3 weeks then every 3 weeks or more frequently as needed
Dose limiting toxicity determination | Weekly assessment for the first 3 weeks
Pharmacokinetic profile evaluation | Day 1 and Day 15

SECONDARY OUTCOMES:
Preliminary tumor response | Every 6 week

CONTACTS AND LOCATIONS:
Overall Officials: Susumu Matsuki, BS, Study Director — Abbott Japan Co.,Ltd

REFERENCES:
- [Result] Asahina H, Tamura Y, Nokihara H, Yamamoto N, Seki Y, Shibata T, Goto Y, Tanioka M, Yamada Y, Coates A, Chiu YL, Li X, Pradhan R, Ansell PJ, McKeegan EM, McKee MD, Carlson DM, Tamura T. An open-label, phase 1 study evaluating safety, tolerability, and pharmacokinetics of linifanib (ABT-869) in Japanese patients with solid tumors. Cancer Chemother Pharmacol. 2012 Jun;69(6):1477-86. doi: 10.1007/s00280-012-1846-6. Epub 2012 Mar 2. PMID 22382879